CLINICAL TRIAL: NCT03039673
Title: Efficacy and Safety of Low-dose IL-2 (Ld-IL-2) as a Treg Enhancer for Controlling Neuro-inflammation in Newly Diagnosed Amyotrophic Lateral Sclerosis (ALS) Patients: A Randomized, Double-blind, Placebo- Controlled, Phase-II Proof of Concept/ Proof of Mechanism Clinical Trial
Brief Title: MIROCALS: Modifying Immune Response and OutComes in ALS
Acronym: MIROCALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H2020/PHRC-N/2014/GB-01; 2015-005347-14 (EudraCT Number)
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: interleukin-2; low-dose interleukin-2
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Riluzole; Interleukin-2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose interleukin-2 (Experimental): Patients randomized to this arm will receive subcutaneous injections of low-dose interleukin-2 in addition to oral Riluzole treatment.
  Intervention: Riluzole Intervention: IL-2
  Interventions: Drug: Riluzole; Drug: IL-2
- Placebo (Placebo Comparator): Patients randomized to this arm will receive subcutaneious placebo injections (5% glucose water solution) in addition to oral Riluzole treatment.
  Intervention: Riluzole Intervention: 5% glucose water solution
  Interventions: Drug: Riluzole; Drug: 5% glucose water solution

INTERVENTIONS:
Drug: Riluzole — All patients will be treated with Riluzole for a period of three months prior to final inclusion and randomization. Riluzole treatment will continue throughout the 18 months of follow-up planned for in this protocol.
  Riluzole treatment is part of routine care for patients with ALS.
Drug: IL-2 — The dose of IL-2 to be used in this study will be 2.0 million IU/day.
  Each treatment course will last 5 days (i.e. 1 sub-cutaneous injection per day for 5 consecutive days). The 5-day course will be repeated every 4-weeks over an 18-month treatment period.
  In case of intolerance, a flexible dose-reduction schedule is available.
  Other Names: low dose interleukin-2; ultra low dose interleukin-2
  Arms: low dose interleukin-2
Drug: 5% glucose water solution — The placebo consists of 5% glucose water solution, which is the matrix with which low-dose IL-2 injections are prepared in the experimental arm. Placebo injections are prepared in exactly the same manner as IL-2 injections, just without the IL-2.
  Each treatment course will last 5 days (i.e. 1 sub-cutaneous injection per day for 5 consecutive days). The 5-day course will be repeated every 4-weeks over an 18-month treatment period.
  Arms: Placebo

SUMMARY:
MIROCALS is a phase II study of ld-IL-2 as a therapeutic agent for ALS. A randomized (1:1), placebo-controlled, double-blind, parallel group trial will be carried out to assess ld-IL-2 safety and clinical efficacy on survival and functional decline in newly diagnosed ALS patients treated for 18 months. Randomization will be stratified according to (i) country (n = 2 levels: UK, France) and (ii) site of onset (n= 2 levels: bulbar vs limb onset).

The primary objective to evaluate the clinical efficacy and safety of the experimental drug (ld IL-2) over an 18 months period in order to establish the proof of concept (PoC) that modifying immune responses through the enhancement of regulatory T cells modifies the rate of ALS disease progression.

DETAILED DESCRIPTION:
The secondary objectives of MIROCALS are:

To validate a new phase-II study design to improve the efficiency of drug development in ALS with early determination of drug response using established biomarkers (BMs).

The aims of this new trial design are:

(i) To shorten future trials duration in ALS using an early drug responding surrogate marker of disease activity; (ii) To establish the proof of mechanism (PoM) of the tested drugs; (iii) To identify drug responder status.

Additional exploratory objectives are:

(i) Deep immune & inflammatory phenotyping (ii) Brain biomarkers (iii) Genomics and Transcriptomics

ELIGIBILITY:
Main Inclusion criteria

* Patient is 18 years old and less than 76 years old
* Possible, Probable, Probable laboratory-supported or Definite ALS as defined by El Escorial Revised ALS diagnostic criteria
* Disease duration <= 24 months
* Slow Vital capacity >= 70% of normal
* No prior or present riluzole treatment
* Lumbar punctures accepted by patient and done

Main Exclusion criteria

* Other neurodegenerative disease that could explain signs or symptoms
* Contra indication for lumbar puncture (history of allergy to xylocaine, presence of contra-indicated treatment, or coagulation test abnormality, clinically significant coagulopathy or thrombocytopenia)
* Non authorized treatment
* Other disease or disorders that could preclude functional assessment, or life-threatening disorders
* Any documented, active, past or present, auto-immune disorders except asymptomatic Hashimoto thyroiditis
* Using assisted ventilation
* Feeding through gastrostomy or nasogastric tube
* Women of child-bearing potential or sexually active man without contraception
* Pregnant or breast feeding woman
* Any clinically significant laboratory abnormality (excepting cholesterol, triglyceride, glucose, CK, ferritin)
* History of documented symptomatic and treated asthma within the past 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Time to death from date of randomization to date of death | Month 21
  Time to death from date of randomization to date of death as documented in death certificates, or date of last documented news for patients lost to follow-up, or 640 days for patients who survive more than 640 days (censoring at 640 days). Death certificates are collected by the centre's principal investigator from the City Hall of the patients' home or birth place.

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Leigh, MD, PhD, Principal Investigator — Brighton and Sussex Medical School; Gilbert Bensimon, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (17):
- France (10):
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - HCL - Hôpital Neurologique P. Wertheimer, Lyon
  - APHM - Hôpital de la Timone, Marseille
  - CHRU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nice - Hôpital Pasteur, Nice
  - APHP - Groupe Hospitalier Pitié-Salpetrière, Paris
  - CENTRE HOSPITALIER DE SAINT BRIEUC - Hôpital Yves Le Foll, Saint-Brieuc
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHRU de Tours - Hôpital Bretonneau, Tours
- United Kingdom (7):
  - Trafford Centre for Biomedical Research, Brighton
  - Institute of Neurological Sciences, Queen Elizabeth University Hospital, Glasgow
  - North-East London and Essex MND Regional Care Centre, London
  - King's MND Care and Research Centre, London
  - Centre for Neuromuscular Diseases - National Hospital of Neurology, London
  - Salford Royal NHS Foundation Trust, Neurology Dept, Manchester
  - Sheffield Care and Research Centre, Sheffield

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Bensimon G, Leigh PN, Tree T, Malaspina A, Payan CA, Pham HP, Klaassen P, Shaw PJ, Al Khleifat A, Amador MDM, Attarian S, Bell SM, Beltran S, Bernard E, Camu W, Corcia P, Corvol JC, Couratier P, Danel V, Debs R, Desnuelle C, Dimitriou A, Ealing J, Esselin F, Fleury MC, Gorrie GH, Grapperon AM, Hesters A, Juntas-Morales R, Kolev I, Lautrette G, Le Forestier N, McDermott CJ, Pageot N, Salachas F, Sharma N, Soriani MH, Sreedharan J, Svahn J, Verber N, Verschueren A, Yildiz O, Suehs CM, Saker-Delye S, Muller C, Masseguin C, Hajduchova H, Kirby J, Garlanda C, Locati M, Zetterberg H, Asselain B, Al-Chalabi A; MIROCALS Study Group. Efficacy and safety of low-dose IL-2 as an add-on therapy to riluzole (MIROCALS): a phase 2b, double-blind, randomised, placebo-controlled trial. Lancet. 2025 May 24;405(10492):1837-1850. doi: 10.1016/S0140-6736(25)00262-4. Epub 2025 May 9. PMID 40354799